CLINICAL TRIAL: NCT05579769
Title: A Phase II Pediatric Study of a Graft-VS.-Host Disease (GVHD) Prophylaxis Regimen With no Calcineurin Inhibitors After Day +60 Post First Allogeneic Hematopoietic Cell Transplant for Hematological Malignancies
Brief Title: Pediatric Study of GVHD Ppx w/o Calcineurin Inhibitors After Day60 Post First Allo HSCT for Hematological Malignancies.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left institution
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNI60
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Hematologic Malignancy; Myeloid Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — ruxolitinib; Mesna; Antilymphocyte Serum; thymoglobulin; Cyclosporine; Cyclosporins; Cyclophosphamide; fludarabine; fludarabine phosphate; Methotrexate; Whole-Body Irradiation; Radiotherapy; Busulfan; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Transplant Patients (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: Mesna; Drug: Anti-thymocyte globulin (ATG); Drug: Cyclosporine; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Methotrexate; Radiation: Total Body Irradiation (radiation treatment); Drug: Bone marrow infusion; Drug: Busulfan; Drug: Thiotepa

INTERVENTIONS:
Drug: Ruxolitinib — Day +40 Dosage and Route of Administration-Ruxolitinib tablets should be administered orally BID, approximately every 12 hours, continuously, Oral
  Other Names: (Jakafi®)
Drug: Mesna — Days -3 and -2 Dosage and Route of Administration-Mesna is dosed based on the cyclophosphamide dose and generally administered in fractionated doses at approximately 20% of the total cyclophosphamide dose, Intravenous.
  Other Names: (Mesnex)
Drug: Anti-thymocyte globulin (ATG) — Days -3, -2 and -1 Dosage and Route of Administration-(7 mg/kg total dose); intravenous.
  Other Names: (Thymoglobulin®, rabbit ATG)
Drug: Cyclosporine — Day -1 Dosage and Route of Administration-3 mg/kg; dose will be adjusted to maintain a steady concentration between 250-350 ng/mL or trough concentration between 175-250 ng/mL when transitioned to intermittent dosing.
  Other Names: (Gengraf)
Drug: Cyclophosphamide — Days -3 and -2 Dosage and Route of Administration-60 mg/kg for 2 consecutive days, (120 mg/kg total dose); intravenous.
  Other Names: (Cytoxan)
Drug: Fludarabine — Days -4, -3 and -2 Dosage and Route of Administration-50 mg/m2 daily for 3 consecutive days (150 mg/m2 total dose) intravenous
  Other Names: (Fludara)
Drug: Methotrexate — Days +1, +3, +6 and +11 Dosage and Route of Administration-10 mg/m2/dose, intravenous
  Other Names: MTX; Amethopterin
Radiation: Total Body Irradiation (radiation treatment) — Days -7, -6, -5 and -4 6.2.3 Target Dose 1200 cGy total dose delivered 150 cGy per treatment fraction delivered BID over 4 days with 6 MV photons.
  Dose rate should be < 10 cGy/min in patients treated at extended SSD (450-500 cm) in the TBI couch and will be less than 15 cGy/min in young children and infants treated at extended SSD (200-220 cm) on the floor.
  Intra-fraction interval should be 6 hours. Custom posteriorly placed (PA only) partial transmission lung shields (blocks) will be used to reduce the average dose to the lung to approximately 1000 cGy total dose.
  An additional 400 cGy supplemental testicular radiation delivered in 2 fractions of 200 cGy delivered for males with lymphoid lineage leukemia.
  Other Names: TBI
Drug: Bone marrow infusion — Day 0
Drug: Busulfan — Days -4, -3 and -2 Dosage and Route of Administration-3.2 mg/kg/day; intravenous.
  Other Names: Busulfex)
Drug: Thiotepa — Days -6 and -5 Dosage and Route of Administration-(10 mg/kg total dose); intravenous
  Other Names: Triplex by Immunex; TESPA; TSPA

SUMMARY:
The participants are being asked to take part in this clinical trial because the participant have a lymphoid or myeloid based cancer diagnosis that requires a bone marrow transplant.

Primary Objectives

To estimate the incidence of severe acute GVHD (saGVHD) using a prophylaxis regimen with no calcineurin inhibitors after day +60 post first allogeneic Human Leukocyte antigen (HLA)-matched sibling or unrelated donor HCT for hematological malignancies.

Secondary objective

Determine the cumulative incidence of relapse, NRM, chronic GVHD, and OS in study participants at one year post-transplant.

Exploratory objectives

* To evaluate the pharmacokinetic/pharmacodynamic (PK/PD) profiles of ruxolitinib, fludarabine, and rATG.
* To assess immune reconstitution in study participants within the first year post-HCT.

DETAILED DESCRIPTION:
The investigator propose to employ two preparative regimens based on the underlying hematological malignancy. For hematological malignancies of the lymphoid lineage we will use a standard preparative regimen consisting of Total Body Irradiation and cyclophosphamide (TBI/Cy), unless TBI is contraindicated. For myeloid malignancies we will use thiotepa, busulfan, and fludarabine (TBF), a preparative regimen that has been associated with a reduced risk of relapse and trend for improved survival with comparable NRM in comparison to busulfan and cyclophosphamide (BuCy), our current regimen. All HCT recipients will receive cyclosporine in combination with methotrexate and ruxolitinib as GVHD prophylaxis. Recipients of MUD HCT will receive rATG for additional immunosuppression as is standard for unrelated donor transplants

ELIGIBILITY:
Inclusion criteria

Diagnosis:

* Patients with high risk acute lymphoblastic leukemia in first remission. Examples include, but are not limited to, patients with certain leukemic cell cytogenetic findings (e.g. t(9;22) or t(4;11)); delayed response to induction chemotherapy; re-emergence of leukemic blasts by MRD (at any level) in patients previously MRD negative; persistently detectable MRD at lower levels; early T-cell precursor (ETP) ALL.
* Patients with acute lymphoblastic leukemia beyond first remission.
* Patients with Hodgkin's disease beyond first remission or with refractory disease.
* Patients with chronic myelogenous leukemia.
* Patients with primary or secondary myelodysplastic syndrome.
* Patients with Non-Hodgkin's lymphoma beyond first remission or with refractory disease.
* Patients with de novo acute myeloid leukemia in or beyond first remission or with relapsed or refractory disease, or myeloid sarcoma (extra-medullary AML).
* Patients with secondary acute myeloid leukemia.
* NK cell lymphoblastic leukemia in any CR.
* Biphenotypic, bilineage, or undifferentiated leukemia.
* Juvenile Myelomonocytic Leukemia (JMML)
* All patients with prior evidence of CNS leukemia must be treated and be in CNS CR.

Patients must have a related or unrelated donor matched at 12 of 12 HLA alleles.

Patient must have a Karnofsky/Lansky score of 70 or higher.

Patients must be 12 years of age or older.

Patients must have a shortening fraction >26% or left ventricular ejection fraction >40%.

Patients must have bilirubin less than or equal to 2.5 mg/dL and alanine aminotransferase (ALT) less than or equal to 5 times the upper limit of normal.

Patients must have creatinine clearance, or a glomerular filtration rate (GFR), greater than 70 mL/min/1.73m2.

Patients must be free of severe infection that upon determination of principal investigator precludes BMT.

Patients must have FVC >50% predicted OR, if unable to perform pulmonary function testing, must maintain pulse oximetry oxygen saturation >92% on room air.

Female patients of childbearing age must have a negative pregnancy test.

Exclusion criteria

* Patients who have undergone prior HCT.
* Patients who have a peripheral blood stem cell graft source.
* Patients who have a non-permissive mismatch at the DPB1 allele.
* Patients who are HIV positive.
* Patients positive for Hepatitis B surface antigen (HBsAg).
* Patients positive for Hepatitis C.
* Patients with latent tuberculosis with positive TB IFN gamma release assay.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Srinivasan, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Body Irradiation (TBI)/Cyclophosphamide (Cy): Patients with lymphoid malignancies will receive Total Body Irradiation (TBI)/Cyclophosphamide (Cy).
  Bone marrow grafts will be used. HLA-identical sibling donors will be considered first followed by histocompatible relatives or unrelated donors. Permissive DPB1 mismatched grafts will be included. Unrelated grafts will be obtained through NMDP or other registries.
  Participants receive 8 doses TBI. Cyclophosphamide, IV. Rabbit ATG, IV. Males with lymphoid lineage leukemia will receive an additional testicular boost concurrent with TBI.
  Patients who receive a bone marrow product from MSD will not receive rATG.
  G-CSF: Use of GCSF is not recommended except after day +21 when a single dose not exceeding 2.5mcg/kg may be given after rounding off if APC is >500 cells/mm3, and ANC is<500 cells/mm3 to mobilize cells.
  Mesna: Mesna will be given IV approximately 15 minutes prior to each dose of cyclophosphamide and approximately 3, 6, 9, and 12 hours after each dose of cyclophosphamide.
  GVHD prophylaxis: Cyclosporine, IV. Methotrexate, IV. Ruxolitinib, Oral or NG.
- Thiotepa, Busulfan, and Fludarabine (TBF): Patients with myeloid, bi-phenotypic, bilineage or undifferentiated leukemia will receive thiotepa, busulfan, and fludarabine (TBF). Patients will receive TBF regimen when TBI is not appropriate.
  Bone marrow grafts will be used. HLA-identical sibling donors will be considered first followed by histocompatible relatives or unrelated donors. Permissive DPB1 mismatched grafts will be included. Unrelated grafts will be obtained through NMDP or other registries.
  Participants receive Thiotepa, IV. Busulfan, IV. Fludarabine, IV. Rabbit ATG, IV.
  Patients who receive a bone marrow product from MSD will not receive rATG.
  G-CSF: Use of GCSF is not recommended except after day +21 when a single dose not exceeding 2.5mcg/kg may be given after rounding off if APC is >500 cells/mm3, and ANC is<500 cells/mm3 to mobilize cells.
  Levetiracetam IV will be prescribed as seizure prophylaxis for recipients receiving busulfan.
  GVHD prophylaxis: Cyclosporine, IV. Methotrexate, IV. Ruxolitinib, Oral or NG.
Period: Overall Study
Arm/Group | Total Body Irradiation (TBI)/Cyclophosphamide (Cy) | Thiotepa, Busulfan, and Fludarabine (TBF)
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants meeting eligibility criteria and who completed study therapy: Allogeneic Human Leukocyte antigen (HLA)-matched sibling or unrelated donor hematopoietic cell transplant (MSD/MUD HCT) for hematological malignancies. Hematological malignancies of the lymphoid lineage will use a standard preparative regimen consisting of Total Body Irradiation and cyclophosphamide (TBI/Cy), unless TBI is contraindicated. Myeloid malignancies will use thiotepa, busulfan, and fludarabine (TBF) regimen.
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Body Irradiation (TBI)/Cyclophosphamide (Cy) | Thiotepa, Busulfan, and Fludarabine (TBF) | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (4.95) | 17 (0) | 16.25 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of saGVHD Using a ProphylaxisRegimen With no Calcineurin Inhibitors After Day 100 Post First Allogeneic HLA-Matched Sibling or Unrelated Donor HCT for Hematological Malignancies.
Description: Development of Severe Acute GVHD (saGVHD) at or before Day 100 post transplant is considered as an event. Severe acute GVHD is defined as grade II-IVGVHD. Acute graft-vs-host disease will be evaluated using the standard grading criteria.
Time Frame: 100 days post transplant
Population: None of the 3 participants had saGVHD.
Measure: Count of Participants; unit: Participants
Groups:
- Total Body Irradiation (TBI)/Cyclophosphamide (Cy): Patients with lymphoid malignancies will receive Total Body Irradiation (TBI)/Cyclophosphamide (Cy).
  Bone marrow grafts will be used. HLA-identical sibling donors will be considered first followed by histocompatible relatives or unrelated donors. Permissive DPB1 mismatched grafts will be included. Unrelated grafts will be obtained through NMDP or other registries.
  TBI/Cy regimen: Participants receive TBI. Cyclophosphamide, IV. Rabbit ATG, IV. Males with lymphoid lineage leukemia will receive an additional testicular boost concurrent with TBI.
  Patients who receive a bone marrow product from MSD will not receive Rabbit ATG.
  G-CSF: Use of GCSF is not recommended unless patients have not engrafted on day +21.
  Mesna: MESNA will be given for bladder protection to patients who receive Cyclophosphamide.
  Levetiracetam IV will be prescribed as seizure prophylaxis for recipients receiving busulfan.
  GVHD prophylaxis: Cyclosporine, IV. Methotrexate, IV. Ruxolitinib, Oral or NG.
- Thiotepa, Busulfan, and Fludarabine (TBF): Patients with myeloid, bi-phenotypic, bilineage or undifferentiated leukemia will receive thiotepa, busulfan, and fludarabine (TBF). Patients will receive TBF regimen when TBI is not appropriate.
  Bone marrow grafts will be used. HLA-identical sibling donors will be considered first followed by histocompatible relatives or unrelated donors. Permissive DPB1 mismatched grafts will be included. Unrelated grafts will be obtained through NMDP or other registries.
  TBF regimen: Thiotepa, IV. Busulfan, IV. Fludarabine, IV. Rabbit ATG, IV.
  Patients who receive a bone marrow product from MSD will not receive Rabbit ATG.
  G-CSF: Use of GCSF is not recommended unless patients have not engrafted on day +21.
  Mesna: MESNA will be given for bladder protection to patients who receive Cyclophosphamide.
  Levetiracetam IV will be prescribed as seizure prophylaxis for recipients receiving busulfan.
  GVHD prophylaxis: Cyclosporine, IV. Methotrexate, IV. Ruxolitinib, Oral or NG.
Arm/Group | Total Body Irradiation (TBI)/Cyclophosphamide (Cy) | Thiotepa, Busulfan, and Fludarabine (TBF)
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

2. Secondary Outcome: Cumulative Incidence of Overall Survival (OS)
Description: The one-year survival is defined by the participant who has not died within one year after post transplantation. The rate is calculated by computing the ratio between total number of one year survival patients and the total number of patients.
Time Frame: One-year post-transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Body Irradiation (TBI)/Cyclophosphamide (Cy) | Thiotepa, Busulfan, and Fludarabine (TBF)
Number analyzed (Participants) | 2 | 1
Participants | 1 | 1

3. Secondary Outcome: Cumulative Incidence of Relapse
Description: Bone marrow studies for disease status evaluation will be performed at 1-year post-transplant. Testing will include a research evaluation for minimal residual disease.
Time Frame: One-year post-transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Body Irradiation (TBI)/Cyclophosphamide (Cy) | Thiotepa, Busulfan, and Fludarabine (TBF)
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

4. Secondary Outcome: Cumulative Incidence of Non Relapse Mortality (NRM)
Description: Non-relapse mortality is death without evidence of disease relapse or progression. The rate is calculated by computing the ratio between total number of NRM patients and the total number of patients.
Time Frame: One-year post-transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Body Irradiation (TBI)/Cyclophosphamide (Cy) | Thiotepa, Busulfan, and Fludarabine (TBF)
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

5. Secondary Outcome: Cumulative Incidence of Chronic GVHD
Description: Chronic graft-vs-host disease will be evaluated using the standard grading criteria.
Time Frame: One-year post-transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Body Irradiation (TBI)/Cyclophosphamide (Cy) | Thiotepa, Busulfan, and Fludarabine (TBF)
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Transplant recipients will be followed for adverse events from the start of conditioning and throughout the first year post-transplant
Description: Recipient participants were followed for all NCI Grade III-V adverse events from the start of conditioning through the first-year post HCT, up to 14 months, regardless of their relationship to the treatment given.
Groups:
- TBI/Cy Regimen: Patients with lymphoid malignancies will receive Total Body Irradiation (TBI)/Cyclophosphamide (Cy).
  Bone marrow grafts will be used. HLA-identical sibling donors will be considered first followed by histocompatible relatives or unrelated donors. Permissive DPB1 mismatched grafts will be included. Unrelated grafts will be obtained through NMDP or other registries.
  Participants receive 8 doses TBI. Cyclophosphamide, IV. Rabbit ATG, IV. Males with lymphoid lineage leukemia will receive an additional testicular boost concurrent with TBI.
  Patients who receive a bone marrow product from MSD will not receive rATG.
  G-CSF: Use of GCSF is not recommended except after day +21 when a single dose not exceeding 2.5mcg/kg may be given after rounding off if APC is >500 cells/mm3, and ANC is<500 cells/mm3 to mobilize cells.
  Mesna: Mesna will be given IV approximately 15 minutes prior to each dose of cyclophosphamide and approximately 3, 6, 9, and 12 hours after each dose of cyclophosphamide.
  GVHD prophylaxis: Cyclosporine, IV. Methotrexate, IV. Ruxolitinib, Oral or NG.
- TBF Regimen: Patients with myeloid, bi-phenotypic, bilineage or undifferentiated leukemia will receive thiotepa, busulfan, and fludarabine (TBF). Patients will receive TBF regimen when TBI is not appropriate.
  Bone marrow grafts will be used. HLA-identical sibling donors will be considered first followed by histocompatible relatives or unrelated donors. Permissive DPB1 mismatched grafts will be included. Unrelated grafts will be obtained through NMDP or other registries.
  Participants receive Thiotepa, IV. Busulfan, IV. Fludarabine, IV. Rabbit ATG, IV.
  Patients who receive a bone marrow product from MSD will not receive rATG.
  G-CSF: Use of GCSF is not recommended except after day +21 when a single dose not exceeding 2.5mcg/kg may be given after rounding off if APC is >500 cells/mm3, and ANC is<500 cells/mm3 to mobilize cells.
  Levetiracetam IV will be prescribed as seizure prophylaxis for recipients receiving busulfan.
  GVHD prophylaxis: Cyclosporine, IV. Methotrexate, IV. Ruxolitinib, Oral or NG.
Arm/Group | TBI/Cy Regimen | TBF Regimen
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI/Cy Regimen (N=2) | TBF Regimen (N=1)
Fever (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Disseminated Adenovirus) (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TBI/Cy Regimen (N=2) | TBF Regimen (N=1)
Blood and lymphatic system disorders - Other, specify (Thrombotic Microangiopathy) (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr virus infection reactivation (Infections and infestations) | 2 (2) | 1 (1)
Fungemia (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcus (Infections and infestations) | 1 (1) | 0 (0) — Upper respiratory infection
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-paukar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic (Vascular disorders) | 1 (1) | 0 (0)
Rhinovirus (Infections and infestations) | 1 (1) | 0 (0) — Upper respiratory infection
Human parainfluenza virus (Infections and infestations) | 1 (1) | 0 (0) — Upper respiratory infection
Rhino/Enterovirus (Infections and infestations) | 1 (1) | 0 (0) — Upper respiratory infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT05579769/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT05579769/ICF_001.pdf